CLINICAL TRIAL: NCT00001986
Title: Double-Blind, Placebo-Controlled, Single-Dose Trial of 1-Octanol in Essential Tremor
Brief Title: 1-Octanol to Treat Essential Tremor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000062; 00-N-0062
Record Dates: First submitted 2000-01-28; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Essential Tremor
Keywords: Alcohol; Octanol; Treatment; Tremor
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — 1-Octanol

INTERVENTIONS:
Drug: 1-Octanol

SUMMARY:
This study will evaluate the safety and effectiveness of the food additive 1-octanol for treating essential tremor. This disorder, which is an involuntary shaking, usually of the hands, has no satisfactory treatment. It affects more than one of every 100 people in the general population, with the figure climbing to nearly 4 in every hundred among people over 40 years old. In animal studies, 1-octanol reduced chemically induced tremors in rats. This study will test the effects of the accepted daily intake of 1-octanol (1 milligram per kilogram of body weight) on essential tremor in humans.

Patients with essential tremor 21 years old and older who wish to enroll in this study will undergo eligibility screening with a medical history and physical examination that includes tests for thyroid, liver and kidney problems. Participants will be randomly assigned to receive either 1-octanol or a placebo (an inactive substance). Patients in both groups will have an intravenous catheter (a thin, plastic tube) placed in an arm vein for collecting blood samples during the study. Those in the 1-octanol group will be given a 1-octanol capsule; the placebo group will receive a look-alike capsule containing no active ingredient. Neither the patient nor the doctor will know which patients are taking 1-octanol or placebo until the end of the study.

Tremors will be measured once before the catheter is placed, every 15 minutes during the first 2 hours after taking the capsule, twice during the third hour (30 minutes apart), and once again after 5 hours. The tremors are measured using procedures called accelerometry and surface electromyography. For these procedures, electrodes are taped to the skin; needles are not used. Blood samples will be collected once before taking the capsule, every 15 minutes for the first hour and a half after taking the capsule and again at 2 hours, 4 hours and 5 hours after taking the capsule. Vital signs (blood pressure, pulse, and respiratory rate) will be measured every 15 minutes during the first 2 hours of taking the capsule, every 30 minutes during the third hour, and again at 4 hours and 5 hours.

Participants will stay in the hospital overnight for observation and return after 3 days for a follow-up physical examination, including a blood test.

DETAILED DESCRIPTION:
Essential tremor (ET) is the most common movement disorder; however, there is currently no satisfactory drug treatment. The neural mechanisms underlying ET remain unknown. One of the prevalent hypotheses is that ET is a result of a defective mechanism that normally dampens the natural oscillations of inferior olive (IO) neurons whose intrinsic oscillatory activity is attributed to the presence of low threshold calcium channels (LTCC). 1-Octanol is known to inhibit LTCC of olivary neurons and was found to reduce the tremor induced in rats with harmaline, an alkaloid known to hyperpolarize IO neurons increasing their tendency to fire rhythmically at rest. The aim of this study is to assess the effects of 1-octanol on ET in humans. This study is designed as a double-blind, placebo-controlled, single-dose trial in untreated patients with ET. Electromyography (EMG) and acclerometry are used to assess tremor before and after 1-octanol administration. The accepted daily intake (ADI) of 1-octanol (1 mg/kg/d) as a food additive will be given as a single dose. Toxicity from octanol will be monitored clinically and by liver function and electrolyte measurements.

ELIGIBILITY:
Patients with essential tremor affecting the upper limbs who are 21 years of age or older.

Patients who are not taking medications for essential tremor or any other medical condition for at least 2 weeks.

Patients who have not consumed alcohol or cold medications containing alcohol for at least 24 hours prior to the day of the study.

Women must not be pregnant or lactating. Women of childbearing age must use birth control while participating in this study.

Patients must not have any neurological disease other than tremor (e.g., Parkinson's disease).

Patients must not have evidence of thyroid, liver, kidney or chronic lung disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2000-01; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bal T, McCormick DA. Synchronized oscillations in the inferior olive are controlled by the hyperpolarization-activated cation current I(h). J Neurophysiol. 1997 Jun;77(6):3145-56. doi: 10.1152/jn.1997.77.6.3145. PMID 9212264
- [Background] Elble RJ. Animal models of action tremor. Mov Disord. 1998;13 Suppl 3:35-9. doi: 10.1002/mds.870131306. PMID 9827592